CLINICAL TRIAL: NCT00150436
Title: An Open-Label Extension Safety and Efficacy Study of Pregabalin in Patients With Postherpetic Neuralgia
Brief Title: To Evaluate Long-Term Safety and Efficacy of Pregabalin in Patients With Postherpetic Neuralgia.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1008-198
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2006-12-22 (Estimated); Status verified 2006-12

CONDITIONS: Neuralgia
MeSH Terms: conditions — Neuralgia | interventions — Pregabalin

INTERVENTIONS:
Drug: Pregabalin

SUMMARY:
To evaluate long-term safety and efficacy of pregabalin in patients with postherpetic neuralgia.

ELIGIBILITY:
Inclusion Criteria:

* Must have met the inclusion criteria for preceding double-blind BID study in postherpetic neuralgia
* Must have received pregabalin/placebo under double-blind conditions for a minimum of 3 weeks.

Exclusion Criteria:

* Patients cannot participate if they experienced a serious adverse event during preceding double-blind BID study which was determined to be related to the study medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276
Dates: Start 2002-02; Study Completion 2005-07

PRIMARY OUTCOMES:
Safety Efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer